CLINICAL TRIAL: NCT06624306
Title: Comparing Efficacy and Complication Between Prone Versus Prone-Flexed Position for Percutaneous Nephrolithotomy (PCNL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Hesham Abdel Azim El Helaly, Assistant Professor, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PF-PCNL
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2023-12

CONDITIONS: Urolithiasis; Kidney Stone; Complication
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- prone PNL (Active Comparator): Prone PNL
  Interventions: Procedure: Prone PNL
- prone-flexed PNL (Active Comparator): prone-flexed PNL
  Interventions: Procedure: Prone-flexed PNL

INTERVENTIONS:
Procedure: Prone PNL — Prone PNL
  Arms: prone PNL
Procedure: Prone-flexed PNL — Prone-flexed PNL
  Arms: prone-flexed PNL

SUMMARY:
Comparing Efficacy and Complication Between Prone Versus Prone-Flexed Position For Percutaneous Nephrolithotomy (PCNL)

ELIGIBILITY:
Inclusion Criteria:

1. Staghorn calculi
2. Renal pelvis stones >2 cm
3. Lower pole stones >1.5 cm
4. SWL-resistant stones

Exclusion Criteria:

1. Age <18 years or Pregnancy
2. Bilateral simultaneous PCNL
3. Need for 3 percutaneous tracts intraoperative
4. Morbid obesity (BMI >40)
5. Non opaque renal stones.
6. Refuse to complete study requirements
7. Atypical bowel interposition need CT guided puncture
8. Tumour in the presumptive access tract area or Potential malignant kidney tumour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparing the prone with the prone-flexed position for PCNL reporting complications | 1 year
  Outcome measures by using the clavien dindo classification system

SECONDARY OUTCOMES:
Assessment of stone free rate of the two groups | 1 year
  Outcome measures by stone fragment residual ≤ 2 mm by computed tomography (CT)

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum faculty of Medicine, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided